CLINICAL TRIAL: NCT03643328
Title: Ex Vivo Evaluation of Immunity Activation Face to Staphylococcus Aureus Antigens and Adjuvants of a Vaccine Candidate in Cells From Haemodialysis Patients
Brief Title: Ex Vivo Evaluation of Immunity Activation Face to S. Aureus Antigens and Adjuvants of a Vaccine Candidate in Cells From Haemodialysis Patients
Acronym: ANTISTAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1608178; ANSM (Other: 2017-A00707-46)
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Staphylococcus Aureus
Keywords: Staphylococcus Aureus; haemodialysis; vaccine; immune response
MeSH Terms: conditions — Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- new haemodialysis patients. (Experimental): There is an analyse of immune response against S. aureus from new haemodialysis patients by blood samples and nasal swabs.
  Interventions: Biological: blood samples; Biological: nasal swabs

INTERVENTIONS:
Biological: blood samples — Blood samples will be collected at inclusion, at 6 months and 12 months for hematological and immunological analyses.
Biological: nasal swabs — Two nasal swabs will be collected at inclusion, at 6 months and 12 months for virology analyses.

SUMMARY:
S. aureus is a leading cause of severe infections notably in haemodialysis patients. These patients have a high risk of S. aureus nasal carriage, with a rate of persistent carriage near 30%. These carriers are particularly at risk of S. aureus infections as we previously shown. High risk of S. aureus infections such as bacteremia occurred notably in patients with dialysis catheters. Decolonization of carriers may prevent such infections however this approach has limits. Development of an effective S. aureus vaccine is crucial. To date, past vaccines tested (phase III) failed to achieve their end points. Target of only one or few antigens, absence of cellular response induction and possibly no impact on carriage are probably the reasons of the failures.

DETAILED DESCRIPTION:
In an attempt to minimize failure in a clinical phase, ex vivo analysis of immune response of leucocytes of haemodialysis patients face to S. aureus and the impact of antigens and adjuvants of a candidate vaccine may help.

ELIGIBILITY:
Inclusion Criteria:

* Patient starting haemodialysis for chronic hemodialysis.
* Patient starting haemodialysis on catheter
* Patient who signed the informed consent form

Exclusion Criteria:

* Pregnant woman
* Patient who starts Haemodialysis for over 3 months
* Patient with anemia (hemoglobin <7 g / dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
EX VIVO measure of innate immunity: functional capacity of neutrophils to S. aureus vaccine antigens | Up to 12 months
  Measured by blood samples at 0, 6 and 12 months
EX VIVO measure of innate immunity: induction of oxidative burst to S. aureus vaccine antigens | Up to 12 months
  Measured by blood samples 0, 6 and 12 months
EX VIVO measure of innate immunity : phenotype activation of different cell types from PBMCs (peripheral blood mononuclear cells) to S. aureus vaccine antigens | Up to 12 months
  Measured by blood samples 0, 6 and 12 months.
EX VIVO measures of innate immunity: chemokines and cytokines secretions to S. aureus vaccine antigens | Up to 12 months
  Measured by blood samples 0, 6 and 12 months.
EX VIVO measure of acquired immunity: measures of S. aureus antibodies titre in serum to S. aureus vaccine antigens | Up to 12 months
  Measured by blood samples 0, 6 and 12 months.

SECONDARY OUTCOMES:
Incidence of persistant portage of S. aureus in the nose haemodialysis patients. | Months 0 and 6 and 12
  Measured by nasal swabs.
Analysis of the S. aureus clonal complexes of nasal carriage strains from haemodialysis patients. | Months 0 and 6 and 12
  Measured by nasal swabs.
Number of infection by S. aureus in new haemodialysis patients. | Month 12
  By data collection
EX VIVO measure of innate immunity: functional capacity of neutrophils to S. aureus vaccine adjuvants | Months 0 and 6 and 12
  Measured by blood samples.
EX VIVO measure of innate immunity: induction of oxidative burst to S. aureus vaccine adjuvants | Months 0 and 6 and 12
  Measured by blood samples.
EX VIVO measure of innate immunity : phenotype activation of different cell types from PBMCs (peripheral blood mononuclear cells) to S. aureus vaccine adjuvants | Months 0 and 6 and 12
  Measured by blood samples.
EX VIVO measures of innate immunity: chemokines and cytokines secretions to S. aureus vaccine adjuvants | Months 0 and 6 and 12
  Measured by blood samples.
EX VIVO measure of acquired immunity: measures of S. aureus antibodies titre in serum to S. aureus vaccine adjuvants | Months 0 and 6 and 12
  Measured by blood samples.
Investigation of the presence of antigens of interest selected for the vaccine approach in strains of S. aureus in the nasal carriage | Months 0 and 6 and 12
  Measured by nasal swabs.
Survival rate to S.aureus in the whole blood | Months 0 and 6 and 12
  Measured by blood samples. Expressed in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth BOTELHO-NEVERS, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No